CLINICAL TRIAL: NCT00412529
Title: A Randomized, Open-label, Controlled, Multicenter, Exploratory Trial to Characterize the Results of Daily Oral Administration of Telbivudine (LDT600) 600 mg or Entecavir (ETV) 0.5 mg Given Over 12 Weeks on the Kinetics of Hepatitis B Virus (HBV) DNA in Adults With HBeAg-positive, Compensated Chronic Hepatitis B (CHB)
Brief Title: Viral Kinetics Study of Telbivudine and Entecavir in Adults With Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600A2407
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-02

CONDITIONS: Hepatitis B; Chronic Hepatitis B
Keywords: HBeAg-positive, chronic hepatitis B; telbivudine; entecavir; viral kinetics
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — entecavir; Telbivudine

ARMS (2):
- Telbivudine (Experimental)
  Interventions: Drug: Telbivudine
- Entecavir (Active Comparator)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Entecavir 0.5 mg once daily for 12 weeks.
  Arms: Entecavir
Drug: Telbivudine — Telbivudine 600 mg once daily for 12 weeks.
  Arms: Telbivudine

SUMMARY:
This exploratory study is designed to determine the early viral kinetic profile during treatment with telbivudine or entecavir at multiple time points over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-70 years of age with documented compensated hepatitis B "e" antigen (HBeAg)-positive chronic hepatitis B
* Able to comply with study regimen and provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Unwilling to use double barrier method of contraception
* Co-infected with hepatitis C virus (HCV), hepatitis D virus (HDV) or human immunodeficiency virus (HIV)
* Received Hepatitis B therapy in the past
* Use of immunomodulatory therapy in past 12 months
* History of or symptoms of hepatic decompensation or pancreatitis
* Frequent or prolonged use of potentially hepatotoxic or nephrotoxic drugs
* Concurrent medication likely to preclude compliance with schedule of evaluations
* Use of other investigational drugs within 30 days of enrollment
* Abnormal laboratory values during screening

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- South Korea (8):
  - Holy Family Hospital_Bucheon, Bucheon,Kyunggi
  - Inje University Busan Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Gachon Univ. Gil Medical Center Hospital, Incheon
  - Asan Medical Center, Seoul
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Medical Center_Anam, Seoul
  - The Catholic University of Korea, Seoul

REFERENCES:
- [Result] Suh DJ, Um SH, Herrmann E, Kim JH, Lee YS, Lee HJ, Lee MS, Lee YJ, Bao W, Lopez P, Lee HC, Avila C, Zeuzem S. Early viral kinetics of telbivudine and entecavir: results of a 12-week randomized exploratory study with patients with HBeAg-positive chronic hepatitis B. Antimicrob Agents Chemother. 2010 Mar;54(3):1242-7. doi: 10.1128/AAC.01163-09. Epub 2009 Dec 22. PMID 20028815
- See also: Early Viral Kinetics of Telbivudine and Entecavir: Results of a 12-Week Randomized Exploratory Study with Patients with HBeAg-Positive Chronic Hepatitis B — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2826006/?tool=pubmed

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telbivudine | Entecavir
Started | 23 | 21
Completed | 23 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telbivudine | Entecavir | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline Measures based on Intention to treat population.
  Years | 36.2 (9.62) | 33.4 (8.82) | 34.9 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Hepatitis B Virus (HBV) DNA Levels
Description: Baseline HBV DNA is defined as the last pre-dose assessment of HBV DNA.
Time Frame: Baseline (day 1) to Week 12 (day 85)
Population: Intent to Treat (ITT) population included all patients who received at least one dose of study drug and had at least one post-baseline assessment of serum HBV DNA. The randomized treatment was used in the analyses of this population.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Telbivudine | Entecavir
Number analyzed (Participants) | 23 | 21
log10 copies/mL
  Baseline (day 1) | 10.290 (1.6477) | 9.721 (1.7141)
  At Week 12 | 3.669 (0.8817) | 3.194 (1.1729)
  Change from Baseline to week 12 | -6.621 (1.5610) | -6.527 (1.5365)

2. Secondary Outcome: Change in Mean HBV DNA Level
Description: Baseline HBV DNA is defined as the last pre-dose assessment of HBV DNA.HBV DNA reductions, considered as the repeated measures, from baseline to Weeks 2, 4, 8.
Time Frame: Baseline (day 1) to Weeks 2, 4, 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Telbivudine | Entecavir
Number analyzed (Participants) | 23 | 21
log10 copies/mL
  Change from Baseline to week 2 :(N=20, 21) | -3.999 (1.3917) [3.04 to 4.30] | -3.974 (1.3460) [3.32 to 4.58]
  Change from Baseline to week 4 : (N= 23, 21) | -5.273 (1.3071) [4.55 to 5.58] | -4.875 (1.5781) [4.58 to 5.61]
  Change from Baseline to week 8 : (N= 23, 21) | -6.161 (1.4937) [5.23 to 6.26] | -5.976 (1.5288) [5.44 to 6.5]

3. Secondary Outcome: The Area Under the Curve (AUC) of HBV DNA Change.
Description: In AUC efficacy analyses, all the visits from baseline to Week 12 visit (including the planned and the repeated) with a non-missing HBV DNA level were included.
Time Frame: From Baseline to Week 12
Population: Intention-to-treat (ITT) population included all patients who received at least one dose of study drug and had at least one post-baseline assessment of serum HBV DNA. The randomized treatment was used in the analyses of this population.
Measure: Mean (Standard Deviation); unit: (log10 copies/mL) * days
Arm/Group | Telbivudine | Entecavir
Number analyzed (Participants) | 23 | 21
(log10 copies/mL) * days | -453.5 (103.13) [369.5 to 462.42] | -442.6 (131.30) [395.87 to 488.79]

4. Secondary Outcome: Change in Alanine Aminotransferase (ALT) Levels
Time Frame: From Baseline to Week 12
Population: Intention to treat (ITT) population included all patients who received at least one dose of study drug and had at least one post-baseline assessment of serum HBV DNA. The randomized treatment was used in the analyses of this population.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Telbivudine | Entecavir
Number analyzed (Participants) | 23 | 21
IU/L
  Baseline | 163.1 (125.29) | 170.2 (152.74)
  At Week 12 | 55.1 (63.92) | 54.0 (36.92)
  Change from Baseline to Week 12 | -108.0 (147.87) | -116.3 (162.81)

5. Secondary Outcome: Characterization of Very Early Viral Kinetics: Estimation of Viral Clearance
Description: Viral kinetic parameters were estimated with a bi-phasic mathematical model:
  V(t) = (1-ε)pI(t) - cV(t)
  I(t) = (1- η)TV(t) - δI(t)
  V serum viral load, I productively infected cells, ε efficiency factor of blocking virus production, p viral production rate, c viral clearance rate, η efficiency factor of blocking de novo infection, β de novo infection rate, T uninfected target cells, δ rate of infected cell loss. Maximum-likelihood estimation for the viral kinetic parameters entailed fitting a nonlinear differential equation system via the least-squares approach from serum HBV DNA data.
Time Frame: Baseline to 12 weeks
Population: Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: clearance per day
Arm/Group | Telbivudine | Entecavir
Number analyzed (Participants) | 23 | 21
clearance per day | 0.809 (0.3904) | 1.002 (0.8162)

6. Secondary Outcome: Characterization of Very Early Viral Kinetics: Estimation of the Rate of Infected Cell Loss
Description: as for outcome 5
Time Frame: Baseline to 12 weeks
Population: Intent to Treat (ITT) population. The value for the rate of infected cell loss for 1 patient in telbivudine arm was not used in calculation of summary statistics for this variable as this patient showed a deviation from the biphasic pattern in viral kinetic modeling.
Measure: Mean (Standard Deviation); unit: infected cell loss per day
Arm/Group | Telbivudine | Entecavir
Number analyzed (Participants) | 22 | 21
infected cell loss per day | 0.075 (0.0231) | 0.071 (0.0227)

7. Secondary Outcome: Characterization of Very Early Viral Kinetics: Estimation of the Efficiency Factor of Blocking Virus Production
Description: Viral kinetic parameters were estimated with a bi-phasic mathematical model of HBV DNA by using compartments of free virus, infected cells, and uninfected target cells. The model parameter of interest was the effectiveness of the drug in blocking virus production from infected cells (efficacy, ε). Blocking efficiency was within the range between 0 and 1.
Time Frame: Baseline to 12 weeks
Population: Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: percentage of blocking efficiency
Arm/Group | Telbivudine | Entecavir
Number analyzed (Participants) | 23 | 21
percentage of blocking efficiency | 0.991 (0.0133) | 0.992 (0.0090)

8. Secondary Outcome: Number of Patients Who Are Polymerase Chain Reaction (PCR) Negative
Description: PCR negative was considered <300 copies/mL. PCR positive was considered =>300 copies/mL.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telbivudine | Entecavir
Number analyzed (Participants) | 23 | 21
Participants
  <300 copies/mL | 2 | 6
  >= 300 copies/mL | 21 | 15

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety population included all patients who received at least one dose of study drug and had at least one post-baseline safety assessment (i.e., adverse event or laboratory assessment).
Arm/Group | Telbivudine | Entecavir
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/21
Other Adverse Events (participants affected / at risk) | 4/23 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telbivudine (N=23) | Entecavir (N=21)
Chest discomfort (General disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telbivudine (N=23) | Entecavir (N=21)
Nausea (Gastrointestinal disorders) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 3 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.